CLINICAL TRIAL: NCT05737654
Title: The Effect of Exercise with Augmented Reality Glasses on Metabolic Parameters, Anthropometric Measurement Values and Quality of Life in Children Aged 10-12 with Type 1 Diabetes
Brief Title: The Effect of Exercise on Metabolic Parameters, Anthropometric Measurement Values and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Harun Özbey, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2022/540
Record Dates: First submitted 2023-01-23; First posted 2023-02-21 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2023-12

CONDITIONS: Type1diabetes; Metabolic Syndrome; Nursing Caries
Keywords: Child with Type 1 Diabetes; Metabolic Parameters; Augmented Reality Glasses; Quality of Life; Anthropometric Values
MeSH Terms: conditions — Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Augmented reality glasses group (Experimental): Two days a week (12 weeks in total), each session will be 60 minutes in total, and moderate exercise will be done with AR glasses.
  Interventions: Other: Exercise with augmented reality glasses
- Control group (No Intervention): No intervention/application will be made to the children who will be included in the control group.

INTERVENTIONS:
Other: Exercise with augmented reality glasses — Two days a week (12 weeks in total), each session will be 60 minutes in total, and moderate exercise will be done with AR glasses.
  Arms: Augmented reality glasses group

SUMMARY:
This study was planned as a randomized controlled experimental study to determine the effect of exercise with Augmented Reality Glasses (AR) on metabolic parameters, anthropometric measurement values and quality of life in children with T1DM aged 10-12 years. The research will be carried out with children aged 10-12 with T1DM who are followed up in Erciyes University Health Application and Research Center Fevzi Mercan-Mustafa Eraslan Children's Hospital Pediatric Endocrinology Outpatient Clinic. A total of 30 (AR exercise group=15 and control group=15) children with T1DM between the ages of 10-12 will be included in the sample of the study, according to the sampling calculation. The data of the study, Descriptive Characteristics Form for Children with T1DM and Their Families, Serum and Urine Biochemistry Values Form, Anthropometric Measurement Values Form, Quality of Life Scale for Children with Diabetes Mellitus Child and Parent Form (PedsQL 3.0), Augmented Reality Glasses, Continuous Glucose Tracker, Blood Glucose Meter, Body Composition Analyzer, Caliper, Tape Measure and Digital Height and Weight Meter. Ethics committee approval from "Erciyes University Clinical Research Ethics Committee" and institutional permission from "ERU Health Application and Research Center Mustafa Eraslan Fevzi Mercan Children's Hospital" were obtained in order to conduct the study. Hypothesis tests, correlation and regression analyzes will be applied according to the suitability of the data for normal distribution. As a result of the study; Exercise practice with augmented reality glasses is expected to improve metabolic parameters and anthropometric measurement values and increase the quality of life in children with T1DM.

The main question it aims to answer are:

Exercise with augmented reality glasses in children with T1DM;

* It has an effect on metabolic parameters.
* It has an effect on anthropometric measurement values.
* It has an effect on the scores of the Quality of Life in Children with Diabetes Mellitus Scale-Child and Parent Form (PedsQL 3.0).

DETAILED DESCRIPTION:
Type 1 Diabetes Mellitus (T1DM) is a chronic metabolic disease characterized by insulin deficiency. T1DM is one of the most common chronic diseases in childhood. In the 10th Diabetes Atlas (2021) data of the International Diabetes Association (IDF), it is stated that the population of children aged 19 and under is 2.61 billion in the world, approximately 1.2 million of these children have T1DM, and there are approximately 150 thousand new children diagnosed with T1DM every year in the world. In the same report, it was stated that there are approximately 26 thousand children aged 19 and under with T1DM in Turkey. T1DM, whose treatment and management is complex, causes both children and their parents to encounter many problems. These problems cause deterioration in quality of life and perceived well-being in children with T1DM. The problems experienced in this direction, adaptation problems and decreased quality of life lead to deterioration of metabolic control in children with T1DM. Children with T1DM who cannot adapt to their disease may have acute and chronic complications that lead to deterioration of metabolic control. One of the most important complications seen in children with T1DM is osteopenia, which tends to increase gradually. Proper nutrition, physical activity, insulin therapy and follow-up of complications have an important place in preventing complications that may develop in children with T1DM, ensuring metabolic control and increasing their quality of life. Exercise in T1DM; reducing the need for insulin and increasing its effect, providing blood glucose control, increasing muscle strength, providing weight control, increasing body fat and muscle mass, increasing body fluid ratio, increasing bone mineralization, positively affecting the cardiovascular system, reducing blood fats, increasing self-conditioning, It provides many benefits such as increasing confidence and reducing stress. Despite the numerous benefits of exercise, studies have shown that children with T1DM do not exercise regularly and do not want to do traditional (walking, running, cycling, swimming, etc.) exercises. In this direction, exercise that requires continuity in diabetes management can be made dynamic for children with T1DM by using different approaches. For this reason, it is thought that structured exercise with augmented reality glasses (AR) that can respond to the reactions of the child with T1DM will be more dynamic and will prevent macrovascular complications such as osteopenia and increase the quality of life in children with T1DM by providing metabolic control.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 10-12,
* Having been diagnosed with Type 1 Diabetes (T1DM) at least six months ago,
* Do not have any other chronic disease other than T1DM,
* No psychiatric diagnosis
* No orthopedic problems,
* Able to read and write
* Can speak Turkish,
* No mental, physical or neurological disability,
* residing in the province where the research will be conducted,
* Children and children with parental consent to participate in the study will be included in the study.

Exclusion Criteria:

* Not showing up on one of the planned workout days,
* Developing unexpected complications (hypoglycemia, hyperglycemia, diabetic ketoacidosis…) during exercise,
* Using another exercise method during the research process,
* Serum and urine biochemistry values cannot be measured,
* Anthropometric measurement values cannot be obtained,
* Have not had their main meal at least three hours before the scheduled exercise time,
* Children who do not have snacks and additional insulin on the planned exercise day will be excluded from the study.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels | Change in average HbA1c levels over 12-week sessions
  HbA1c levels of children with type 1 diabetes before, during, after exercise and during the control session.
Change in body mass index | Change in average body mass index over 12-week sessions
  Average body mass index values of children with type 1 diabetes before, during, after exercise and during the control session.
Change in quality of life | Change in average quality of life values over 12-week sessions
  Quality of life scale in children with Type 1 Diabetes Mellitus (PedsQL 3.0) Varni et al. (2003) developed by This scale measures both general areas of quality of life and disease-specific areas. The scale is a comprehensive, multidimensional scale made with both diabetic children and surrogate (parent/caregiver) notifications. In the scale prepared according to the five-point Likert system, 0 = never creates a problem, 1 = almost never creates a problem, 2 = sometimes creates a problem, 3 = often creates a problem, and 4 = always poses a problem. A linear translation is applied in the total score calculation of the scale and it turns into 0-100 points. The answer to the question is scored 100 if it is marked as never, 75 if it is marked as rarely, 50 if it is marked as sometimes, 25 if it is marked as often, and 0 if it is marked as almost always. The higher the total score, the better the perceived health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Bayat, PhD, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ozbey H, Bayat M. The effect of exercise with augmented reality glasses on metabolic parameters, anthropometric measurement values and quality of life in children aged 10-12 with type 1 diabetes: A randomized controlled trial. J Pediatr Nurs. 2025 Nov-Dec;85:239-248. doi: 10.1016/j.pedn.2025.08.002. Epub 2025 Aug 7. PMID 40780014